CLINICAL TRIAL: NCT05282069
Title: A Multicenter, Double-blind, Placebo-controlled and Active-reference, Randomized, Parallel, Therapeutic Confirmatory Clinical Study to Evaluate the Efficacy and Safety of DA-8010 in Patients With Overactive Bladder
Brief Title: A Study to Evaluate the Efficacy and Safety of DA-8010 in Patients With Overactive Bladder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA8010_OAB_III
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — DA-8010; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): DA-8010 placebo + Solifenacin succinate placebo
  Interventions: Drug: DA-8010 Placebo; Drug: Solifenacin succinate placebo
- DA-8010 2.5mg (Experimental): DA-8010 2.5mg + Solifenacin succinate placebo
  Interventions: Drug: DA-8010 2.5mg; Drug: Solifenacin succinate placebo
- DA-8010 5mg (Experimental): DA-8010 5mg + Solifenacin succinate placebo
  Interventions: Drug: DA-8010 5mg; Drug: Solifenacin succinate placebo
- Solifenacin 5mg (Active Comparator): DA-8010 placebo + Solifenacin succinate 5mg
  Interventions: Drug: DA-8010 Placebo; Drug: Solifenacin 5mg

INTERVENTIONS:
Drug: DA-8010 Placebo — Participants receive placebo to match DA-8010 orally once a day.
  Arms: Placebo; Solifenacin 5mg
Drug: DA-8010 2.5mg — Participants receive DA-8010 2.5mg orally once a day.
  Arms: DA-8010 2.5mg
Drug: DA-8010 5mg — Participants receive DA-8010 5mg orally once a day.
  Arms: DA-8010 5mg
Drug: Solifenacin 5mg — Participants receive solifenacin 5 mg orally once a day.
  Arms: Solifenacin 5mg
Drug: Solifenacin succinate placebo — Participants receive placebo to match solifenacin 5 mg orally once a day.
  Arms: DA-8010 2.5mg; DA-8010 5mg; Placebo

SUMMARY:
This study will evaluate the efficacy and safety of DA-8010 in patients with overactive bladder for 12 weeks as double-blind, placebo-controlled and active-reference study, and also will evaluate the long-term safety of DA-8010 for 52 weeks in patients with overactive bladder as open-label study.

ELIGIBILITY:
Inclusion Criteria:

Main Inclusion at Screening (Visit 1):

* Men and women 19 years or older with OAB symptoms for ≥ 3 months.
* Subject who is willing and able to complete the voiding diary correctly.
* Subject who is willing and able to provide informed consent indicating that they understand the purpose and procedures required for the study

Exclusion Criteria:

Main Exclusion at Screening (Visit 1):

* Clinically significant stress urinary incontinence or mixed urinary incontinence where stress is the predominant factor
* Subject who has Injury or neurodegenerative disease which is able to effect on lower urinary tract and nerves
* Subject with diabetes insipidus, urinary stone, urinary tract infection, interstitial cystitis, recurrent urinary tract infection, pelvic organ prolapse or neurogenic bladder
* Clinically significant benign prostatic hyperplasia at the discretion of the investigator
* Had bladder or lower urinary tract surgery within 12 months from the screening visit
* Medical history of malignant tumor in urinary system or pelvic organs
* >150 mL of post-void residual volume in the screening test

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the mean number of micturitions per 24 hours at 12 weeks | 12 weeks
  Change from baseline in the mean number of micturitions per 24 hours at 12 weeks

SECONDARY OUTCOMES:
Change from baseline in the mean number of micturitions per 24 hours at 4 and 8 weeks | 4 and 8 weeks
  Change from baseline in the mean number of micturitions per 24 hours at 4 and 8 weeks
Change from baseline in the mean number of urinary urgency(Grade 2, 3, 4) per 24 hours at 4, 8 and 12 weeks | 4, 8 and 12 weeks
  Change from baseline in the mean number of urinary urgency(Grade 2, 3, 4) per 24 hours at 4, 8 and 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes